CLINICAL TRIAL: NCT03863145
Title: Open Label, Multicenter, Phase 1 Study to Evaluate the Maximum Tolerated Dose of Orally Administered CB-03-10 With Dose Expansion Phase, in Subjects With Advanced Solid Tumors
Brief Title: Study to Evaluate Maximum Tolerated Dose of Oral CB-03-10 With Dose Expansion Phase, in Advanced Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cosmo Technologies Ltd (Industry)
Responsible Party: Sponsor
Organization: Cosmo Pharmaceuticals NV (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CB-03-10/01
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Advanced Refractory Solid Tumors; Subjects Considered Likely to Respond to CB-03-10

STUDY DESIGN:
Intervention Model Description: Part 1 (Dose Escalation): Subjects with advanced refractory solid tumors Part 2 (Dose Expansion): Defined subject subgroups considered likely to respond to CB-03-10 (eg, relapsed/refractory pancreatic adenocarcinoma, androgen independent prostate adenocarcinoma, triple-negative breast adenocarcinoma) or indications that demonstrated activity in Part 1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Part 1 (Dose Escalation): 100 mg daily.
  Interventions: Drug: CB-03-10

INTERVENTIONS:
Drug: CB-03-10 — CB-03-10, 100 mg capsule for oral use

SUMMARY:
Subjects will undergo baseline evaluation and an assessment of extent of disease.

Subjects in Part 1 (Dose Escalation) will receive escalating doses of CB-03-10 based on a modified Fibonacci schema using a standard oncology 3+3 study design to define an MTD and a RP2D. Plasma PK samples will be collected at predetermined timepoints for all subjects.

Subjects in Part 2 (Dose Expansion) of the study will receive CB-03-10 at the RP2D determined in the Part 1 of the study. The indications included in each group will be determined at the completion of Part 1 of the study by Safety Review Committee (SRC).

Subjects will be evaluated weekly initially (for 2 cycles in Part 1 and for 1 cycle in Part 2) and every 2 weeks thereafter. Reassessment of disease will be conducted at Week 8 and every 8 weeks thereafter. Subjects with evidence of response (partial or complete) will be re-evaluated at least 4 weeks later for confirmation.

DETAILED DESCRIPTION:
Subjects will undergo baseline evaluation and an assessment of extent of disease.

Subjects in Part 1 (Dose Escalation) will receive escalating doses of CB-03-10 based on a modified Fibonacci schema using a standard oncology 3+3 study design to define an MTD and a RP2D. Plasma PK samples will be collected at predetermined timepoints for all subjects.

Subjects in Part 2 (Dose Expansion) of the study will receive CB-03-10 at the RP2D determined in the Part 1 of the study. The indications included in each group will be determined at the completion of Part 1 of the study by Safety Review Committee (SRC).

Subjects will be evaluated weekly initially (for 2 cycles in Part 1 and for 1 cycle in Part 2) and every 2 weeks thereafter. Reassessment of disease will be conducted at Week 8 and every 8 weeks thereafter. Subjects with evidence of response (partial or complete) will be re-evaluated at least 4 weeks later for confirmation.

ELIGIBILITY:
INCLUSION CRITERIA:

Signed informed consent For Part 1 (Dose Escalation): Histologically or cytologically confirmed relapsed or refractory locally advanced or metastatic solid tumor, not amenable to standard therapy For Part 2 (Dose Expansion): Histologically or cytologically confirmed relapsed or refractory locally advanced or metastatic solid tumor limited to a specific tumor subtype as determined by the SRC Age >18 years Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 For Part 1 (Dose Escalation): Measurable or evaluable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) criteria For Part 2 (Dose Expansion): Measurable disease as per RECIST v1.1 criteria. Adequate renal, hepatic and bone marrow function as defined by Screening labs Negative pregnancy test for females of childbearing potential at the Screening Visit and use of appropriate method of birth control.

EXCLUSION CRITERIA Pregnant or breastfeeding women Known central nervous system (CNS) metastases or spinal cord compression Known second cancer of other primary origin (excluding Stage I non-melanoma skin cancer and prostate cancer controlled with hormonal therapy) within the prior 5 years Active autoimmune disease Significant cardiac disease Uncontrolled hypertension Major surgery or irradiation within 28 days prior to start of study treatment Fewer than 28 days (or fewer than 5 half-lives, whichever is shorter) from prior anticancer therapy Requirement for chronic corticosteroids or other immunosuppressant drugs Known infection with hepatitis B or C virus Known infection with HIV and CD4+ T-cell counts < 350 cells/uL Patients with an opportunistic infection within the past 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose | 29 days
  Determine the maximum tolerated dose (MTD) of CB-03-10 in subjects with advanced solid tumors
Determine the dose-limiting toxicity | 28 days
  Determine the dose-limiting toxicity (DLT) of CB-03-10 in subjects with advanced solid tumors

SECONDARY OUTCOMES:
Determine a recommended Phase 2 dose (RP2D) of CB-03-10 | 28 days
  Determine a recommended Phase 2 dose (RP2D) of CB-03-10

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California Irvine Health Chao Family Comprehensive Cancer Center, California City, California
  - University of Colorado Cancer Center, Colorado Springs, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Barbara Ann Karmanos Cancer Institute, Michigan Center, Michigan
  - Gabrail Cancer Center, Ohio City, Ohio
  - Tranquil Clinical Research, Texas City, Texas

REFERENCES:
- [Result] Fleming TR. One-sample multiple testing procedure for phase II clinical trials. Biometrics. 1982 Mar;38(1):143-51. PMID 7082756
- [Result] Von Hoff DD, Ramanathan RK, Borad MJ, Laheru DA, Smith LS, Wood TE, Korn RL, Desai N, Trieu V, Iglesias JL, Zhang H, Soon-Shiong P, Shi T, Rajeshkumar NV, Maitra A, Hidalgo M. Gemcitabine plus nab-paclitaxel is an active regimen in patients with advanced pancreatic cancer: a phase I/II trial. J Clin Oncol. 2011 Dec 1;29(34):4548-54. doi: 10.1200/JCO.2011.36.5742. Epub 2011 Oct 3. PMID 21969517
- [Result] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Result] Conroy T, Gavoille C, Samalin E, Ychou M, Ducreux M. The role of the FOLFIRINOX regimen for advanced pancreatic cancer. Curr Oncol Rep. 2013 Apr;15(2):182-9. doi: 10.1007/s11912-012-0290-4. PMID 23341367
- [Result] Brower V. New approaches tackle rising pancreatic cancer rates. J Natl Cancer Inst. 2014 Dec 22;106(12):dju417. doi: 10.1093/jnci/dju417. Print 2014 Dec. No abstract available. PMID 25535299
- [Result] Schweizer MT, Gulati R, Mostaghel EA, Nelson PS, Montgomery RB, Yu EY, Cheng HH. Docetaxel-related toxicity in metastatic hormone-sensitive and metastatic castration-resistant prostate cancer. Med Oncol. 2016 Jul;33(7):77. doi: 10.1007/s12032-016-0793-1. Epub 2016 Jun 14. PMID 27300548
- [Result] Block TS, Murphy TI, Munster PN, Nguyen DP, Lynch FJ. Glucocorticoid receptor expression in 20 solid tumor types using immunohistochemistry assay. Cancer Manag Res. 2017 Mar 6;9:65-72. doi: 10.2147/CMAR.S124475. eCollection 2017. PMID 28293120
- [Result] Stringer-Reasor EM, Baker GM, Skor MN, Kocherginsky M, Lengyel E, Fleming GF, Conzen SD. Glucocorticoid receptor activation inhibits chemotherapy-induced cell death in high-grade serous ovarian carcinoma. Gynecol Oncol. 2015 Sep;138(3):656-62. doi: 10.1016/j.ygyno.2015.06.033. Epub 2015 Jun 24. PMID 26115975
- [Result] Pan D, Kocherginsky M, Conzen SD. Activation of the glucocorticoid receptor is associated with poor prognosis in estrogen receptor-negative breast cancer. Cancer Res. 2011 Oct 15;71(20):6360-70. doi: 10.1158/0008-5472.CAN-11-0362. Epub 2011 Aug 25. PMID 21868756
- [Result] Wu W, Chaudhuri S, Brickley DR, Pang D, Karrison T, Conzen SD. Microarray analysis reveals glucocorticoid-regulated survival genes that are associated with inhibition of apoptosis in breast epithelial cells. Cancer Res. 2004 Mar 1;64(5):1757-64. doi: 10.1158/0008-5472.can-03-2546. PMID 14996737
- [Result] Kach J, Long TM, Selman P, Tonsing-Carter EY, Bacalao MA, Lastra RR, de Wet L, Comiskey S, Gillard M, VanOpstall C, West DC, Chan WC, Griend DV, Conzen SD, Szmulewitz RZ. Selective Glucocorticoid Receptor Modulators (SGRMs) Delay Castrate-Resistant Prostate Cancer Growth. Mol Cancer Ther. 2017 Aug;16(8):1680-1692. doi: 10.1158/1535-7163.MCT-16-0923. Epub 2017 Apr 20. PMID 28428441
- [Result] Kroon J, Puhr M, Buijs JT, van der Horst G, Hemmer DM, Marijt KA, Hwang MS, Masood M, Grimm S, Storm G, Metselaar JM, Meijer OC, Culig Z, van der Pluijm G. Glucocorticoid receptor antagonism reverts docetaxel resistance in human prostate cancer. Endocr Relat Cancer. 2016 Jan;23(1):35-45. doi: 10.1530/ERC-15-0343. Epub 2015 Oct 19. PMID 26483423
- [Result] Yemelyanov A, Bhalla P, Yang X, Ugolkov A, Iwadate K, Karseladze A, Budunova I. Differential targeting of androgen and glucocorticoid receptors induces ER stress and apoptosis in prostate cancer cells: a novel therapeutic modality. Cell Cycle. 2012 Jan 15;11(2):395-406. doi: 10.4161/cc.11.2.18945. Epub 2012 Jan 15. PMID 22223138
- [Result] Szmulewitz RZ, Chung E, Al-Ahmadie H, Daniel S, Kocherginsky M, Razmaria A, Zagaja GP, Brendler CB, Stadler WM, Conzen SD. Serum/glucocorticoid-regulated kinase 1 expression in primary human prostate cancers. Prostate. 2012 Feb 1;72(2):157-64. doi: 10.1002/pros.21416. Epub 2011 May 11. PMID 21563193
- [Result] Puhr M, Hoefer J, Eigentler A, Ploner C, Handle F, Schaefer G, Kroon J, Leo A, Heidegger I, Eder I, Culig Z, Van der Pluijm G, Klocker H. The Glucocorticoid Receptor Is a Key Player for Prostate Cancer Cell Survival and a Target for Improved Antiandrogen Therapy. Clin Cancer Res. 2018 Feb 15;24(4):927-938. doi: 10.1158/1078-0432.CCR-17-0989. Epub 2017 Nov 20. PMID 29158269
- [Result] Isikbay M, Otto K, Kregel S, Kach J, Cai Y, Vander Griend DJ, Conzen SD, Szmulewitz RZ. Glucocorticoid receptor activity contributes to resistance to androgen-targeted therapy in prostate cancer. Horm Cancer. 2014 Apr;5(2):72-89. doi: 10.1007/s12672-014-0173-2. Epub 2014 Mar 11. PMID 24615402
- [Result] Arora VK, Schenkein E, Murali R, Subudhi SK, Wongvipat J, Balbas MD, Shah N, Cai L, Efstathiou E, Logothetis C, Zheng D, Sawyers CL. Glucocorticoid receptor confers resistance to antiandrogens by bypassing androgen receptor blockade. Cell. 2013 Dec 5;155(6):1309-22. doi: 10.1016/j.cell.2013.11.012. PMID 24315100
- [Result] Schweizer MT, Yu EY. Persistent androgen receptor addiction in castration-resistant prostate cancer. J Hematol Oncol. 2015 Nov 13;8:128. doi: 10.1186/s13045-015-0225-2. PMID 26566796
- [Result] Traina TA, Miller K, Yardley DA, Eakle J, Schwartzberg LS, O'Shaughnessy J, Gradishar W, Schmid P, Winer E, Kelly C, Nanda R, Gucalp A, Awada A, Garcia-Estevez L, Trudeau ME, Steinberg J, Uppal H, Tudor IC, Peterson A, Cortes J. Enzalutamide for the Treatment of Androgen Receptor-Expressing Triple-Negative Breast Cancer. J Clin Oncol. 2018 Mar 20;36(9):884-890. doi: 10.1200/JCO.2016.71.3495. Epub 2018 Jan 26. PMID 29373071
- [Result] Munoz J, Wheler JJ, Kurzrock R. Androgen receptors beyond prostate cancer: an old marker as a new target. Oncotarget. 2015 Jan 20;6(2):592-603. doi: 10.18632/oncotarget.2831. PMID 25595907
- [Result] Robinson-Rechavi M, Escriva Garcia H, Laudet V. The nuclear receptor superfamily. J Cell Sci. 2003 Feb 15;116(Pt 4):585-6. doi: 10.1242/jcs.00247. No abstract available. PMID 12538758
- [Result] Stringer EM, Saha P, Swoboda A, Kocherginsky M, Baker G, Olberkyte S, et al. A phase I trial of mifepristone (M), carboplatin (C), and gemcitabine (G) in advanced breast and ovarian cancer. J Clin Oncol. 2017;35 (15 sup(1083):1083.
- See also: National Cancer Institute. Cancer of the Esophagus - SEER Stat Fact Sheets [Internet]. Cancer Statistics. 2015 [cited 2015 Sep 15]. — http://seer.cancer.gov/statfacts/html/esoph.html
- See also: International Council on Harmonisation. Addendum to ICH E11: Clinical Investigation of Medicinal Products in the Pediatric Population e11(r1). Vol. Step 4, ICH Harmonised Guideline E11 (R1). 2017. — https://www.ich.org/fileadmin/Public_Web_Site/ICH_Products/Guidelines/Efficacy/E11/E11-R1EWG_Step4_Addendum_2017_0818.pdf
- See also: International Conference on Harmonization Guidance on Good Clinical Practice [Internet]. [cited 2016 Jan 1]. — http://www.ich.org/home.html